CLINICAL TRIAL: NCT06470087
Title: A Randomized Controlled Clinical Trial Comparing High Purity Type-I Collagen-based Skin Substitute to Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers
Brief Title: High Purity Type I Collagen Based Skin Substitute Vs Dehydrated Human Amnion/Chorion Membrane in Treatment of DFUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Principal Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor & HoD, Department of Plastic Reconstructive & Aesthetic Surgery, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPTC101
Record Dates: First submitted 2024-05-31; First posted 2024-06-24 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer (DFU)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SOC and Type-I Collagen-based Skin Substitute (Other): Arm 1 -The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Interventions: Device: SOC and Type-I Collagen-based Skin Substitute
- SOC and Human Amnion/Chorion Membrane (Other): Arm 2: The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Interventions: Other: SOC and Human Amnion/Chorion Membrane

INTERVENTIONS:
Device: SOC and Type-I Collagen-based Skin Substitute — Arm 1 -The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Arms: SOC and Type-I Collagen-based Skin Substitute
Other: SOC and Human Amnion/Chorion Membrane — Arm 2: The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous paraffin gauze (Cuticel), second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap (Crepe Bandage)
  Arms: SOC and Human Amnion/Chorion Membrane

SUMMARY:
This is a randomized controlled clinical investigation in patients suffering from diabetic foot ulcers. The study intends to compare patient outcome data using Standard of Care with Type-I Collagen-based Skin Substitute and Standard of Care with Dehydrated Human Amnion/Chorion Membrane.

DETAILED DESCRIPTION:
The purpose of this randomized controlled clinical study is to collect and compare patient outcome data at 4 weeks using Type-I Collagen-based Skin Substitute in one half of the patients and Dehydrated Human Amnion/Chorion Membrane in the other half.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age or older.
* Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At randomization subjects must have a target diabetic foot ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 10.0 cm2 measured post debridement using a ruler to measure wound area.
* The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
* The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
* The target ulcer must be full thickness on the foot or ankle that does not probe to bone.
* Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

  * Transcutaneous Oxygen Measurement (TCOM) ≥30 mmHg
  * Ankle-Brachial Index (ABI) between 0.7 and 1.3
  * Peripheral Vascular Resistance (PVR): Biphasic
  * Toe-Brachial Index (TBI) ˃0.6
  * As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle of the target extremity.
* If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The subject must consent to using the prescribed off-loading method for the duration of the study.
* The subject must agree to attend the twice-weekly/weekly study visits required by the protocol.
* The subject must be willing and able to participate in the informed consent process.
* Patients must have read and signed the IRB approved ICF before screening procedures are undertaken.

Exclusion Criteria:

* A subject known to have a life expectancy of <6 months.
* If the target ulcer is infected or if there is cellulitis in the surrounding skin.
* Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
* A subject that has an infection in the target ulcer that requires systemic antibiotic therapy.
* A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
* Topical application of steroids to the ulcer surface within one month of initial screening.
* A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
* A subject with a glycated hemoglobin (HbA1c) greater than or equal to 13% taken at or within 3 months of the initial screening visit.
* A subject with a serum creatinine ≥ 3.0mg/dL within 6 months of the initial screening visit.

  o A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer.
* Women who are pregnant or considering becoming pregnant within the next 6 months.
* A subject with end stage renal disease requiring dialysis.
* A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
* A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — RajaRajeswari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhanraj P, Naveen N, Babu KR, Mahesh MS, Hanumanthaiah KS. Healicoll: An alternate to flap cover for bare bones and tendons. Acta Medica International. 2016 Jan 1;3(1):146-50
- [Background] Wolfe EM, Mathis SA, de la Olivo Munoz N, Ovadia SA, Panthaki ZJ. Comparison of human amniotic membrane and collagen nerve wraps around sciatic nerve reverse autografts in a rat model. Biomater Biosyst. 2022 Apr 7;6:100048. doi: 10.1016/j.bbiosy.2022.100048. eCollection 2022 Jun. PMID 36824162
- [Background] Mohammed YA, Farouk HK, Gbreel MI, Ali AM, Salah AA, Nourelden AZ, Gawad MMA. Human amniotic membrane products for patients with diabetic foot ulcers. do they help? a systematic review and meta-analysis. J Foot Ankle Res. 2022 Sep 14;15(1):71. doi: 10.1186/s13047-022-00575-y. PMID 36104736
- [Background] DiDomenico LA, Orgill DP, Galiano RD, Serena TE, Carter MJ, Kaufman JP, Young NJ, Jacobs AM, Zelen CM. Use of an aseptically processed, dehydrated human amnion and chorion membrane improves likelihood and rate of healing in chronic diabetic foot ulcers: A prospective, randomised, multi-centre clinical trial in 80 patients. Int Wound J. 2018 Dec;15(6):950-957. doi: 10.1111/iwj.12954. Epub 2018 Jul 17. PMID 30019528
- [Background] Huang Y, Kyriakides TR. The role of extracellular matrix in the pathophysiology of diabetic wounds. Matrix Biol Plus. 2020 Apr 22;6-7:100037. doi: 10.1016/j.mbplus.2020.100037. eCollection 2020 May. PMID 33543031
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (5.98) | 52.3 (7.16) | 50.9 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (2.28) | 25.3 (2.08) | 25.4 (2.11)
Smoking [Count of Participants; unit: Participants]
  Smoking (Present) | 3 | 3 | 6
  Smoking (Absent) | 11 | 11 | 22
Hypertension [Count of Participants; unit: Participants]
  Hypertension (Present) | 2 | 3 | 5
  Hypertension (Absent) | 12 | 11 | 23
Doppler Scan Findings [Count of Participants; unit: Participants]
  Biphasic Flow | 4 | 5 | 9
  Triphasic Flow | 10 | 9 | 19
Glcosylated Hemoglobin [Mean (Standard Deviation); unit: mmol/mol] | 5.8 (0.27) | 5.8 (0.25) | 5.8 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Wound Area Epithelialization From Week 1 Through 4
Description: Percentage wound area epithelialization from week 1 through 4 measured manually with digital photography. Calculated by using:
  Percentage Epithelialization=(Epithelialized Area / Total Wound Area)×100
Time Frame: 4 weeks
Population: The number given indicates the average change in wound area in both the groups between baseline and week 4. Since in all the study participants the wound area has decreased, the value in the table indicates average decrease in wound area in both the groups.
Measure: Mean (Standard Deviation); unit: percentage wound area epithelialization
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
percentage wound area epithelialization | 93.62 (0.12) | 77.71 (0.28)

2. Secondary Outcome: Proportion of Subjects That Obtain Complete Closure Over 4-week Treatment Period
Description: The proportion of subjects that obtain complete closure over the 4-week treatment period
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
Participants | 10 | 7

3. Secondary Outcome: Percenatge of Participants Undergoing Repeat Applications of Advanced Skin Substitute & Human Amnion/Chorion Membrane Used to Obtain Wound Closure
Description: Percenatge of participants undergoing repeat applications of Advanced Skin Substitute & Human Amnion/Chorion Membrane used to obtain wound closure. Since the participants who underwent repeat applications in both groups had only one repeat application, instead of the mean number of repeat applications we are indicating the percentage of participants having repeat applications in both the groups.
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
Participants | 5 | 4

4. Other Pre Specified Outcome: Appearance
Description: Visual observation of the newly formed skin for signs of redness, swelling and other abnormalities.
  Appearance was assessed using visual analog scale, wherein the scale ratings ranged from 0 to 5 where 0 refers to worst appearance and 5 refers to best appearance
Time Frame: The appearance of thewound was assessed only once i.e at the end of 5th week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
units on a scale | 2.5 (0.52) | 2.2 (0.69)

5. Other Pre Specified Outcome: Structural Stability of the Scar
Description: Structural stability of the healed wound will be assessed by compression testing using a blunt-edged tool. Following assessment by the blunt tool, structural stability was rated on 5 point visual anaog scale, where 1 represents fragile and 5 represents stable wound
Time Frame: The appearance of the woundd was assessed only once i.e. at the end of 5th week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
units on a scale | 3.43 (1.02) | 2.71 (0.91)

6. Other Pre Specified Outcome: Wound Recurrence
Description: Subject will be observed for any recurrence of the wound after its closure during the 1-week follow-up
Time Frame: During 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 14 | 14
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 1 month
Description: All the study participants were considered at risk for adverse events. However, no adverse events were observed in the study.
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Small study group. The findings of the study is applicable only to those individuals without any vascular compromise.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT06470087/Prot_SAP_002.pdf